CLINICAL TRIAL: NCT07125859
Title: Prevalence of Preoperative Malnutrition and Changes in Nutritional Status Following Preoperative Nutrition Education in Surgical Patients Attending a Preoperative Clinic
Brief Title: Malnutrition Prevalence and Nutritional Change After Preoperative Nutrition Counseling
Status: Recruiting | Type: Observational
Sponsor: Siriraj Hospital (Other)
Responsible Party: Principal Investigator, Mingkwan Wongyingsinn, MD, Associate Professor, Siriraj Hospital
Other Study IDs: 594/2568 (IRB2)
Record Dates: First submitted 2025-08-04; First posted 2025-08-15 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Nutrition Status
Keywords: Preoperative; Malnutrition; Nutrition education
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Preoperative nutrition risk or Malnutrition is a prevalent up to 65% of surgical patients, leading to significant negative outcomes such as increased complications, poor wound healing, and higher healthcare costs. Preoperative nutrition status is a modifiable risk factor that can be optimized to improve surgical outcomes. Preoperative malnutrition screening creates an opportunity to identify and optimize the nutritional status of at-risk patients before surgery. This study is initiated to determine the prevalence of malnutrition among surgical patients enrolled in an Enhanced recovery after surgery (ERAS) program, using the SPENT and modified Nutrition Alert Form (NAF) during their visit to the preoperative clinic and evaluate the impact of preoperative nutrition education on body weight and nutrition status prior to surgery.

DETAILED DESCRIPTION:
Preoperative nutrition risk or malnutrition negative impacts patients' ability to tolerate surgical stress, impairs wound healing, delays postoperative physical recovery, prolong hospital stay, and increases risk of infection, anemia, impaired gut function, skeletal muscle loss, overall postoperative complications, and healthcare cost.1-6 Importantly, preoperative nutrition status is a modifiable risk factor that can be optimized to improve surgical outcomes.6 However, malnutrition screening is not yet routinely integrated into all surgical pathways.7 Furthermore, only a small proportion of at-risk patients receive preoperative nutrition therapy.7,8 Recent literatures reports that up to 65% of patients admitted for surgery are either malnutrition or at risk of nutrition.7,9-11 This highlights the necessity of preoperative nutrition screening and intervention are needed to enhance postoperative outcomes. The importance of nutritional optimization extends beyond the immediate preoperative period and into the preadmission phase, forming a critical component of the perioperative care continuum, as emphasized by Enhanced Recovery After Surgery (ERAS) guidelines and prehabilitation program.12 Increased awareness has led to several strategies, including preoperative nutrition education, reducing of perioperative fasting, introduction of oral carbohydrate loading before surgery, and early postoperative feeding -all contributing to improved recovery.13,14 Despite growing awareness, considerable variation exists in the tools and criteria used to screen and assess malnutrition, which contributes to inconsistent prevalence data and may hinder timely intervention. Various nutrition screening tools are used worldwide, including the Malnutrition Screening Tool-Short Form (MST-SF), Mini Nutritional Assessment -Short Form (MNA-SF), Nutrition Risk Screening 2002 (NRS-2002), and the Malnutrition Universal Screening Tool (MUST). In Thailand, the SPENT Nutrition Screening Tool, endorsed by the Society of Parenteral and Enteral Nutrition of Thailand (SPENT), is commonly used in clinical settings. For more comprehensive evaluation, nutritional assessment tools such as the Subjective Global Assessment (SGA), Patient-Generated Subjective Global Assessment (PG-SGA), Global Leadership Initiative on Malnutrition (GLIM) criteria, Mini Nutritional Assessment (MNA), and the ASPEN/Academy of Nutrition and Dietetics Malnutrition Indicators (AAIM) are applied internationally. The modified Nutrition Alert Form (NAF), a simplified nutrition assessment tool, is also widely used in Thailand for preoperative patients due to its practicality and ease of use.15-17 This heterogeneity of tools, each incorporating different parameters and thresholds-such as BMI, recent weight loss, dietary intake, and disease burden-results in variability in sensitivity and specificity, complicating comparisons and underscoring the need for standardization tailored to surgical patients.

The reported prevalence of malnutrition in surgical patients varies widely depending on the type of surgery, socioeconomic background, presence of malignancy, and the screening tool used.15 Preoperative malnutrition screening creates an opportunity to identify and optimize the nutritional status of at-risk patients before surgery. Nevertheless, it remains underutilized due to barriers such as time limit and lack of awareness.16,17 The primary aim of this study is to determine the prevalence of malnutrition among surgical patients enrolled in an Enhanced recovery after surgery (ERAS) program, using the SPENT and modified Nutrition Alert Form (NAF) during their visit to the preoperative clinic. The secondary aim is to evaluate the impact of preoperative nutrition education on body weight and nutrition status prior to surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged ≥18 years.
2. Enrolled in the Enhanced Recovery After Surgery (ERAS) program.
3. Referred to the SiPAP program for prehabilitation prior to elective surgery.
4. screened for malnutrition risk using the Society of Parenteral and Enteral Nutrition of Thailand (SPENT) screening tool.
5. Complete clinical records available for analysis.

Exclusion Criteria: Have incomplete nutritional records.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients who enroll to Enhanced Recovery After Surgery (ERAS) program, Siriraj Hospital and referred to the SiPAP program.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
The prevalence of malnutrition using NAF score | Baseline
  The prevalence of malnutrition using Modified Nutrition Alert Form (NAF) score The minimum value for the NAF (Nutritional Assessment Form) is 0 and the maximum value is 88. The NAF uses a combination of BMI, serum albumin or total lymphocyte count to assess nutritional status, with scores ranging from 0-5 (NAF = A, normal to mild malnutrition), 6-10 (NAF = B, moderate malnutrition), and 11 or higher (NAF = C, severe malnutrition).

SECONDARY OUTCOMES:
The change in Modified NAF score | Preoperative period (up to 12 weeks before surgery)
  Changes in Nutrition status measured with change in Modified Modified Nutrition Alert Form (NAF) score. The minimum value for the NAF (Nutritional Assessment Form) is 0 and the maximum value is 88. The NAF uses a combination of BMI, serum albumin or total lymphocyte count to assess nutritional status, with scores ranging from 0-5 (NAF = A, normal to mild malnutrition), 6-10 (NAF = B, moderate malnutrition), and 11 or higher (NAF = C, severe malnutrition).

CONTACTS AND LOCATIONS:
Overall Officials: Mingkwan Wongyingsinn, Principal Investigator — Siriraj Hospital
Locations (1):
- Faculty of Medicine Siriraj Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pischart K, Khemworapong K, Chaopotong P, Achariyapota V. Malnutrition Prevalence and Its Implications on Surgical and Oncological Outcomes in Advanced Ovarian Cancer Patients: A Comprehensive Analysis. Obstet Gynecol Int. 2025 May 10;2025:2918759. doi: 10.1155/ogi/2918759. eCollection 2025. PMID 40384994
- [Background] Chaiwat O, Wongyingsinn M, Muangpaisan W, Chalermsri C, Siriussawakul A, Pramyothin P, Thitisakulchai P, Limpawattana P, Thanakiattiwibun C. A simpler screening tool for sarcopenia in surgical patients. PLoS One. 2021 Sep 23;16(9):e0257672. doi: 10.1371/journal.pone.0257672. eCollection 2021. PMID 34555077
- [Background] Komindrg S, Tangsermwong T, Janepanish P. Simplified malnutrition tool for Thai patients. Asia Pac J Clin Nutr. 2013;22(4):516-21. doi: 10.6133/apjcn.2013.22.4.06. PMID 24231010
- [Background] Karsegard VL, Ferlay O, Maisonneuve N, Kyle UG, Dupertuis YM, Genton L, Pichard C. [Simplified malnutrition screening tool: Malnutrition Universal Screening Tool (MUST)]. Rev Med Suisse Romande. 2004 Oct;124(10):601-5. French. PMID 15573502
- [Background] Grass F, Cerantola Y, Schafer M, Muller S, Demartines N, Hubner M. Perioperative nutrition is still a surgical orphan: results of a Swiss-Austrian survey. Eur J Clin Nutr. 2011 May;65(5):642-7. doi: 10.1038/ejcn.2011.13. Epub 2011 Feb 23. PMID 21346714
- [Background] Higashiguchi T, Arai H, Claytor LH, Kuzuya M, Kotani J, Lee SD, Michel JP, Nogami T, Peng N. Taking action against malnutrition in Asian healthcare settings: an initiative of a Northeast Asia Study Group. Asia Pac J Clin Nutr. 2017 Mar;26(2):202-211. doi: 10.6133/apjcn.022016.04. PMID 28244696
- [Background] Nakahara S, Nguyen DH, Bui AT, Sugiyama M, Ichikawa M, Sakamoto T, Nakamura T. Perioperative nutrition management as an important component of surgical capacity in low- and middle-income countries. Trop Med Int Health. 2017 Jul;22(7):784-796. doi: 10.1111/tmi.12892. Epub 2017 Jun 13. PMID 28510990
- [Background] Gustafsson UO, Scott MJ, Hubner M, Nygren J, Demartines N, Francis N, Rockall TA, Young-Fadok TM, Hill AG, Soop M, de Boer HD, Urman RD, Chang GJ, Fichera A, Kessler H, Grass F, Whang EE, Fawcett WJ, Carli F, Lobo DN, Rollins KE, Balfour A, Baldini G, Riedel B, Ljungqvist O. Guidelines for Perioperative Care in Elective Colorectal Surgery: Enhanced Recovery After Surgery (ERAS(R)) Society Recommendations: 2018. World J Surg. 2019 Mar;43(3):659-695. doi: 10.1007/s00268-018-4844-y. PMID 30426190
- [Background] Weimann A, Braga M, Carli F, Higashiguchi T, Hubner M, Klek S, Laviano A, Ljungqvist O, Lobo DN, Martindale RG, Waitzberg D, Bischoff SC, Singer P. ESPEN practical guideline: Clinical nutrition in surgery. Clin Nutr. 2021 Jul;40(7):4745-4761. doi: 10.1016/j.clnu.2021.03.031. Epub 2021 Apr 19. PMID 34242915
- [Background] Lobo DN, Gianotti L, Adiamah A, Barazzoni R, Deutz NEP, Dhatariya K, Greenhaff PL, Hiesmayr M, Hjort Jakobsen D, Klek S, Krznaric Z, Ljungqvist O, McMillan DC, Rollins KE, Panisic Sekeljic M, Skipworth RJE, Stanga Z, Stockley A, Stockley R, Weimann A. Perioperative nutrition: Recommendations from the ESPEN expert group. Clin Nutr. 2020 Nov;39(11):3211-3227. doi: 10.1016/j.clnu.2020.03.038. Epub 2020 Apr 18. PMID 32362485
- [Background] Ligthart-Melis GC, Luiking YC, Kakourou A, Cederholm T, Maier AB, de van der Schueren MAE. Frailty, Sarcopenia, and Malnutrition Frequently (Co-)occur in Hospitalized Older Adults: A Systematic Review and Meta-analysis. J Am Med Dir Assoc. 2020 Sep;21(9):1216-1228. doi: 10.1016/j.jamda.2020.03.006. Epub 2020 Apr 21. PMID 32327302
- [Background] Geurden B, Franck E, Weyler J, Ysebaert D. The Risk of Malnutrition in Community-Living Elderly on Admission to Hospital for Major Surgery. Acta Chir Belg. 2015 Sep-Oct;115(5):341-7. doi: 10.1080/00015458.2015.11681126. PMID 26560000
- [Background] Bozzetti F, Gianotti L, Braga M, Di Carlo V, Mariani L. Postoperative complications in gastrointestinal cancer patients: the joint role of the nutritional status and the nutritional support. Clin Nutr. 2007 Dec;26(6):698-709. doi: 10.1016/j.clnu.2007.06.009. Epub 2007 Aug 1. PMID 17683831
- [Background] Williams DGA, Ohnuma T, Krishnamoorthy V, Raghunathan K, Sulo S, Cassady BA, Hegazi R, Wischmeyer PE. Postoperative Utilization of Oral Nutrition Supplements in Surgical Patients in US Hospitals. JPEN J Parenter Enteral Nutr. 2021 Mar;45(3):596-606. doi: 10.1002/jpen.1862. Epub 2020 Jun 3. PMID 32492762
- [Background] Wischmeyer PE, Carli F, Evans DC, Guilbert S, Kozar R, Pryor A, Thiele RH, Everett S, Grocott M, Gan TJ, Shaw AD, Thacker JKM, Miller TE, Hedrick TL, McEvoy MD, Mythen MG, Bergamaschi R, Gupta R, Holubar SD, Senagore AJ, Abola RE, Bennett-Guerrero E, Kent ML, Feldman LS, Fiore JF Jr; Perioperative Quality Initiative (POQI) 2 Workgroup. American Society for Enhanced Recovery and Perioperative Quality Initiative Joint Consensus Statement on Nutrition Screening and Therapy Within a Surgical Enhanced Recovery Pathway. Anesth Analg. 2018 Jun;126(6):1883-1895. doi: 10.1213/ANE.0000000000002743. PMID 29369092
- [Background] Prado CM, Ford KL, Gonzalez MC, Murnane LC, Gillis C, Wischmeyer PE, Morrison CA, Lobo DN. Nascent to novel methods to evaluate malnutrition and frailty in the surgical patient. JPEN J Parenter Enteral Nutr. 2023 Feb;47 Suppl 1(Suppl 1):S54-S68. doi: 10.1002/jpen.2420. Epub 2022 Dec 5. PMID 36468288
- [Background] Curtis LJ, Bernier P, Jeejeebhoy K, Allard J, Duerksen D, Gramlich L, Laporte M, Keller HH. Costs of hospital malnutrition. Clin Nutr. 2017 Oct;36(5):1391-1396. doi: 10.1016/j.clnu.2016.09.009. Epub 2016 Sep 19. PMID 27765524
- [Background] Yamamoto T, Shimoyama T, Umegae S, Kotze PG. Impact of Preoperative Nutritional Status on the Incidence Rate of Surgical Complications in Patients With Inflammatory Bowel Disease With Vs Without Preoperative Biologic Therapy: A Case-Control Study. Clin Transl Gastroenterol. 2019 Jun;10(6):e00050. doi: 10.14309/ctg.0000000000000050. PMID 31136361
- [Background] Kim E, Lee DH, Jang JY. Effects of Preoperative Malnutrition on Postoperative Surgical Outcomes and Quality of Life of Elderly Patients with Periampullary Neoplasms: A Single-Center Prospective Cohort Study. Gut Liver. 2019 Nov 15;13(6):690-697. doi: 10.5009/gnl18469. PMID 30970428
- [Background] Wolf JH, Ahuja V, D'Adamo CR, Coleman J, Katlic M, Blumberg D. Preoperative Nutritional Status Predicts Major Morbidity After Primary Rectal Cancer Resection. J Surg Res. 2020 Nov;255:325-331. doi: 10.1016/j.jss.2020.05.081. Epub 2020 Jun 25. PMID 32593891
- [Background] Moon MS, Kim SS, Lee SY, Jeon DJ, Yoon MG, Kim SS, Moon H. Preoperative nutritional status of the surgical patients in Jeju. Clin Orthop Surg. 2014 Sep;6(3):350-7. doi: 10.4055/cios.2014.6.3.350. Epub 2014 Aug 5. PMID 25177463